CLINICAL TRIAL: NCT04687943
Title: Comparison of PELOID Therapy and Kinesio Tape Effectiveness in Patients With Lateral Epicondylitis
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Süleyman Gül, medical doctor, Konya Meram State Hospital
Other Study IDs: KonyaFizikTedaviYazır
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Lateral Epicondylitis; Patient Engagement
MeSH Terms: conditions — Tennis Elbow; Patient Participation | interventions — Mud Therapy; Athletic Tape; Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PELOID therapy: A total of 15 sessions of peloid therapy for 3 weeks, 5 days a week for 42 patients in the first group
  Interventions: Combination Product: PELOID therapy, kinesio tape, exercise
- Kinesio tape: 42 patients in group 2 will be given 2 sessions of muscle and fascia correction techniques per week, with kinesio tape application and cold application
  Interventions: Combination Product: PELOID therapy, kinesio tape, exercise
- Exercise: 42 patients in the third group will be given 3 sets of 10 repetitions home exercise programs for 3 weeks
  Interventions: Combination Product: PELOID therapy, kinesio tape, exercise

INTERVENTIONS:
Combination Product: PELOID therapy, kinesio tape, exercise — 126 patients diagnosed with lateral epicondylitis will be divided into 3 groups. Totally 15 sessions of peloid therapy for 42 patients in 1 group for 3 weeks, 5 days a week, 2 sessions of muscle and fascia correction techniques for 3 weeks in the second group for 3 weeks, and 3 sets per day for 42 patients in the third group for 3 weeks. You will be given 10 repetitive home workouts.

SUMMARY:
In this study, the difference in effectiveness between PELOID therapy and kinesio tape in the treatment of lateral epicondylitis; It was planned to evaluate the effects of these treatments on pain, functionality, activities of daily living and quality of life.

DETAILED DESCRIPTION:
This study was conducted between November 2017 and January 2021 with 126 patients who applied to Konya Training and Research Hospital Physical Therapy and Rehabilitation outpatient clinic with complaints of elbow pain and were diagnosed with lateral epicondylitis, who met the inclusion criteria and did not meet the inclusion criteria.

Lateral epicondylitis diagnosis will be made according to clinical criteria. For the clinical diagnosis of Lateral epicondylitis, if there is resistant wrist extension and pain by pressing the lateral epicondyle of the humerus, Lateral epicondylitis will be diagnosed. Other pathologies that may present with elbow pain will be ruled out. Detailed stories of all participants will be taken and detailed physical examinations will be made. Sociodemographic and clinical characteristics of the participants will be determined by questions such as age, gender, height, weight, educational status, employment status and income level.

126 patients diagnosed with Lateral epicondylitis will be divided into 3 groups. Totally 15 sessions of peloid therapy for 42 patients in 1 group for 3 weeks, 5 days a week, 2 sessions of muscle and fascia correction techniques for 3 weeks in the second group, and 3 sets per day for 42 patients in the third group for 3 weeks. You will be given a home exercise program with 10 repetitions.

In addition, the home exercise program will be shown to both groups. Cold application: At the beginning of each treatment, gel ice packs are wrapped with a moist towel and placed around the elbow joint for 15 minutes. will be applied.

PELOID therapy; PELOIDs are naturally and indigenous to the hot springs; They are used in clinics or packaged at home.In the local peloid application, as the effects of heat; increase in blood flow, decrease in peripheral vein tone, increase in heart rate and heart rate, slight increase in systolic blood pressure, decrease in diastolic pressure, increase in cell division, decrease in viscosity in skin fluids, warm analgesia, increased elasticity in tendons, ligaments and fascia, general sedation, hormonal stimulation (stress hormones, pituitary adrenal cortex and medulla), adaptive effect, elongation of collagen tissue. Vasodilation occurs in the deep parts of the body with the stimulation formed in the parts of the body that come into contact with the peloid, and vasodilation occurs in the deep parts of the body. In addition, hot applications have an anti-inflammatory effect in chronic inflammation. As a result of the studies done, with PELOID therapy; it has positive effects on the symptoms and functional capacity of osteoarthritis; It has significant positive effects on parameters such as the number of painful and swollen joints, morning stiffness, and subjective pain in inflammatory rheumatic diseases; It has been observed that combined therapies are more successful than single treatments, and with the repetition of the treatments, adaptation to work increases, workday loss and treatment costs decrease. Hot peloid is applied to the area as a 1.5-2 cm thick layer. The surface of the application area is covered with a material that provides transparent impermeability, the temperature of the mixture is maintained and it is covered with a towel.

PELOID therapy was applied to our patients at a temperature of 45 degrees for 20 minutes on the elbow. At the end of the application (20 minutes later), the peloid layer is removed and discarded again not to be used. The treatment area is cleaned with soft cloths soaked in hot water. The patient is 10-15 minutes. the session is completed by resting.

Kinesio Taping Application: In addition to classical physiotherapy, kinesio taping was applied to the second group; Lateral epicondylitis taping, consisting of muscle technique and fascia correction techniques, will be performed.Theoretically, it is thought to increase the space between the skin and muscles by raising the skin, relieving this pressure on neural and sensory receptors formed in the tissue due to any reason and supporting the increase of blood and lymph circulation. This effect seen in the circulatory system reduces edema and inflammation and accelerates tissue healing. The reduction in inflammation provides a reduction in pain. Activating the gate control mechanism and the pattern inhibitory mechanisms through mechanoreceptors are also accepted as other mechanisms of pain reduction. When the pain reduction by taping is explained according to the gate control theory; The band reduces the inputs transmitted from the nerve fibers to the nociceptors. Convulsions seen on the skin after tape application raise the skin and reduce painful stimuli by decreasing the pressure on subcutaneous nociceptors. Stretching the skin and applying pressure to the skin stimulate the cutaneous mechanoreceptors. Proprioceptive sensation can be increased by the ability of these mechanoreceptors to change joint motion information.Belt applications can be named as I, Y, X, rake, net or ring depending on their appearance. Type of tape to be applied; It varies according to the technique, the stage of the disease, the length of the muscle, the application area and the targeted treatment. Since I and Y strips are used to reduce pain and edema, they are the most common application methods. Y-strips are also used to surround the muscle to facilitate or suppress movement.

The X-strip method is generally used in cases where the origo and insertion of the muscle changes due to movements or when they are stretched to the maximum, the lengths of which vary greatly and involve the double joint. The rake shape is used especially for reducing edema and for lymph drainage. The web shape created by modifying the rake (fan) shape is used in highly mobile joints such as elbow joints. In order to prevent skin discomfort, the beginning and end regions of the tape should not be stretched during the applications.

Kinesiology tape application is applied with different degrees of tension according to the treatment purpose. The amount of stretching; Maximum stretching (100%), submaximal stretching (75%), moderate stretching (50%), light stretching (25%), very light stretching (10-15%) and no stretching. A total of 6 sessions of kinesio taping will be applied 2 sessions per week. The tapes will remain on the tissue for 48 hours and patients will be asked to remove the tape before coming for treatment.

Home Exercise Program: Patients will be given a home exercise program consisting of eccentric strengthening exercises and stretching exercises, which are planned to increase resistance every week. To the patients; for forearm pronation-supination with wrist extensors Strengthening exercises will be taught and a home exercise program will be started as 3 sets of 10 repetitions per day.

All groups will be evaluated at the beginning of the treatment, in the 3rd week after the treatment and in the 4th week after treatment.

During the evaluations; Pain intensity and pain localization with 0-10 point Visual Analogue Scale (VAS), 0-10 point pain questioning with Visual Analogue Scale (VAS) during one, maximum grip, Arm-Shoulder and Hand Distortion Questionnaire (Arm Disabled, Shoulder and Hand) (DASH) and function and disability, Patient-Rated Forearm Evaluation Questionnaire (PRFEQ) finds the pain and functions of the arm in a 1-week period, and the Short Form-36 (SF-36) will be used in life course. . Visual Analogue Scale (VAS) (0-10 cm); Jamar Hand Dynamometer for pain intensity and pain localization; Visual Analogue Scale (VAS) (0-10 cm) for maximum hand grip strength; Arm-Shoulder and Hand Injury Questionnaire (Arm, Shoulder and Hand Barriers (DASH) Questionnaire) to ensure the level of pain during maximum hand grip; Patient-Based Forearm Assessment Questionnaire (Patient-Graded Forearm Assessment Questionnaire (PRFEQ)) for function and disability; To learn the pain and functions of the arm in a 1-week period, Short Form-36 (SF-36); It has been used for life continues.

ELIGIBILITY:
Inclusion Criteria:

* The patient has pain in the lateral elbow
* Tenderness over the lateral epicondyle
* Pain for at least 3 months with resistant wrist extension
* Between the ages of 18-65

Exclusion Criteria:

* Under the age of 18 or over 65
* Those with communication problems
* Those with a history of injection, surgery, or physical therapy for Lateral epicondylitis within the last 1 year
* Those with a history of cervical and shoulder problems, a history of polyneuropathy, a history of uncontrollable systemic disease (cardiovascular, pulmonary, hepatic, renal, hematologic), those with a history of systemic endocrine disease (DM, Hyperthyroidism)
* Major psychiatric diseases
* Rheumatic diseases such as fibromyalgia, polymyalgia rheumatica, ankylosing spondylitis, rheumatoid arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 126 patients between the ages of 18-65 were included in the study according to the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
PELOID THERAPY AND KINESIO TAPE PROVIDES PAIN REDUCTION IN DAILY LIFE ACTIVITIES OF PATIENTS | November 2017-January 2021
  Significant reduction in VAS pain severity scale is expected in patients with PELOID therapy and kinesio tape application.
PELOID THERAPY AND KINESIO TAPE INCREASES PATIENT'S HAND GRIP | November 2017-January 2021
  After both treatments, there was a significant increase in grip strength evaluated by Jamar dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gul S, Yilmaz H, Karaarslan F. Comparison of the effectiveness of peloid therapy and kinesio taping in tennis elbow patients: a single-blind controlled study. Int J Biometeorol. 2022 Apr;66(4):661-668. doi: 10.1007/s00484-021-02225-7. Epub 2021 Nov 27. PMID 34837528